CLINICAL TRIAL: NCT00556998
Title: An Open-Label, Intravenous To Oral Switch, Multiple Dose Study To Evaluate The Pharmacokinetics, Safety And Tolerability Of Voriconazole In Immunocompromised Adolescents Aged 12 To <17 Years Who Are At High Risk For Systemic Fungal Infection
Brief Title: A Multiple-Dose Study To Evaluate The Pharmacokinetics And Safety Of Voriconazole In Immunocompromised Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: A1501081
Record Dates: First submitted 2007-11-09; First posted 2007-11-12 (Estimated); Results first posted 2012-03-16 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-03

CONDITIONS: Pharmacokinetics
Keywords: pharmacokinetics and safety data of voriconazole in immunocompromised adolescents
MeSH Terms: interventions — Voriconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Voriconazole

INTERVENTIONS:
Drug: Voriconazole — Voriconazole will be used for prophylaxis purpose. 6 mg/kg IV q12h on the first day (Day 1) and 4 mg/kg IV q12h for at least 5.5 days. The IV treatment is no more than 20 days. Then switch to 300 mg oral tablets q12h for at least 6.5 days. The total treatment duration is no more than 30 days.
  Other Names: Vfend

SUMMARY:
This study is designed to collect additional pharmacokinetic and safety data of voriconazole in immunocompromised adolescents receiving intravenous and oral voriconazole. This will help establish voriconazole dosing recommendations for adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are expected to develop neutropenia following chemotherapy.
* Subjects who require treatment for the prevention of systemic fungal infection.

Exclusion Criteria:

* Subjects with a history of severe intolerance of azole antifungal agents.
* Subjects with documented bacterial or viral infection at the time of study entry who are not responding to appropriate treatment against the infection.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2008-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- United States (8):
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Fort Worth, Texas
  - Pfizer Investigational Site, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- All Treatments: Voriconazole intravenous (IV) loading dose (6 mg/kg) was administered in the morning and evening on Day 1, and the IV maintenance dose (4 mg/kg) was administered in the morning and evening on Days 2 to 7 (up to Day 20 if clinically indicated). The oral maintenance dosing regimen (300 mg every 12 hours or 150 mg every 12 hours if subject weighed less than 40 kg) was administered following voriconazole IV and lasted 6.5 days (up to Day 30 if clinically indicated).
Period: Voriconazole Intravenous (IV)
Arm/Group | All Treatments
Started | 26
Treated | 26
Completed | 21 (One participant received 2 days of oral; then received IV again before discontinuing from study.)
Not Completed | 5
Not completed — Adverse Event | 1
Not completed — Other | 4
Period: Voriconazole Oral
Arm/Group | All Treatments
Started | 22 (One participant received voriconazole 150 mg every 12 hours during oral phase.)
Completed | 20
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Intolerant of oral treatment | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Treatments
Number analyzed (Participants) | 26
Age, Customized [Number; unit: Years]
  12 | 4
  13 | 10
  >13 to <17 | 12
Sex/Gender, Customized [Number; unit: Participants]
  Female | 9
  Male | 17

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve Over Dosing Interval at Steady State (AUC12,ss) Following IV Administration
Description: AUC12,ss = Area under the plasma concentration-time profile from time zero (predose) to twelve hours at steady-state. AUC12,ss was obtained by the Linear/Log trapezoidal method.
Time Frame: Day 7 (up to Day 20) at predose, 40, 78 minutes, 4, 6, 8 and 12 hours after start of infusion
Population: Intent to treat (ITT) population of participants who had completed pharmacokinetic (PK) blood sampling for at least one day. N = number of participants with analyzable data.
Measure: Geometric Mean (Standard Deviation); unit: μg*h/mL
Groups:
- Voriconazole IV: Voriconazole IV loading dose (6 mg/kg) in the morning and evening on Day 1 and multiple IV doses (4 mg/kg) in the morning and evening on Days 2 to 7 (up to Day 20 if clinically indicated).
Arm/Group | Voriconazole IV
Number analyzed (Participants) | 23
μg*h/mL | 22.39 (21.47)

2. Primary Outcome: Peak Plasma Concentration at Steady State (Cmax,ss) Following IV Administration
Time Frame: Day 7 (up to Day 20) at predose, 40, 78 minutes, 4, 6, 8 and 12 hours after start of infusion
Population: ITT population of participants who had completed PK blood sampling for at least one day. N = number of participants with analyzable data.
Measure: Geometric Mean (Standard Deviation); unit: μg/mL
Arm/Group | Voriconazole IV
Number analyzed (Participants) | 23
μg/mL | 3.89 (2.59)

3. Primary Outcome: Time to Reach Cmax (Tmax) Following IV Administration
Time Frame: Day 7 (up to Day 20) at predose, 40, 78 minutes, 4, 6, 8 and 12 hours after start of infusion
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Voriconazole IV
Number analyzed (Participants) | 23
hours | 1.30 [1.17 to 3.95]

4. Primary Outcome: AUC12,ss Following Oral Administration
Description: as for outcome 1
Time Frame: Day 7 (up to Day 30) at predose, 1, 2, 4, 6, 8, and 12 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: μg*h/mL
Groups:
- Voriconazole Oral: Oral maintenance dosing regimen (300 mg every 12 hours or 150 mg every 12 hours if subject weighed less than 40 kg) was administered following voriconazole IV and lasted 6.5 days (up to Day 30 if clinically indicated).
Arm/Group | Voriconazole Oral
Number analyzed (Participants) | 19
μg*h/mL | 16.74 (13.50)

5. Primary Outcome: Cmax,ss Following Oral Administration
Time Frame: Day 7 (up to Day 30) at predose, 1, 2, 4, 6, 8, and 12 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: μg/mL
Arm/Group | Voriconazole Oral
Number analyzed (Participants) | 19
μg/mL | 2.35 (1.41)

6. Primary Outcome: Tmax Following Oral Administration
Time Frame: Day 7 (up to Day 30) Predose, 1, 2, 4, 6, 8, and 12 hours postdose
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Voriconazole Oral
Number analyzed (Participants) | 19
hours | 2.00 [0.67 to 8.10]

7. Secondary Outcome: AUC12 Following IV Loading Dose
Description: AUC12 = Area under the plasma concentration-time profile from time zero (predose) to twelve hours. AUC12 was obtained by the Linear/Log trapezoidal method.
Time Frame: Day 1 at predose, 60, 118 minutes, 4, 6, 8 and 12 hours after start of infusion
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: μg*h/mL
Groups:
- Voriconazole IV: Voriconazole IV loading dose (6 mg/kg) in the morning and evening on Day 1.
Arm/Group | Voriconazole IV
Number analyzed (Participants) | 22
μg*h/mL | 9.14 (4.90)

8. Secondary Outcome: Tmax Following an IV Loading Dose
Time Frame: Day 1 at predose, 60, 118 minutes, 4, 6, 8 and 12 hours after start of infusion
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Voriconazole IV
Number analyzed (Participants) | 22
hours | 1.97 [1.90 to 2.08]

9. Secondary Outcome: Cmax Following an IV Loading Dose
Time Frame: Day 1 at predose, 60, 118 minutes, 4, 6, 8 and 12 hours after start of infusion
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: μg/mL
Arm/Group | Voriconazole IV
Number analyzed (Participants) | 22
μg/mL | 2.25 (0.86)

10. Secondary Outcome: Minimum Observed Plasma Trough Concentration (Cmin)
Time Frame: Day 7 (up to Day 20) for IV; Day 7 (up to Day 30) for oral at predose
Population: ITT population of participants who had completed PK blood sampling for at least one day. N = number of participants with analyzable data; n = number of participants who contributed to data.
Measure: Geometric Mean (Standard Deviation); unit: μg/mL
Groups:
- All Treatments: Voriconazole intravenous (IV) loading dose (6 mg/kg) was administered in the morning and evening on Day 1, and the IV maintenance dose (4 mg/kg) was administered in the morning and evening on Days 2-7 (up to Day 20 if clinically indicated). The oral maintenance dosing regimen was administered following voriconazole IV and lasted 6.5 days (up to Day 30 if clinically indicated).
Arm/Group | All Treatments
Number analyzed (Participants) | 21
μg/mL
  IV Day 7 (up to Day 20) (n=21) | 1.05 (1.85)
  Oral Day 7 (up to Day 30) (n=19) | 0.72 (0.81)

11. Secondary Outcome: AUC12,ss of N-oxide Voriconazole Metabolite (UK-121, 265) Following IV Administration
Description: as for outcome 1
Time Frame: Day 1 at predose, 60, 118 minutes, 4, 6, 8 and 12 hours after start of infusion and on Day 7 (up to Day 20) at predose, 40, 78 minutes, 4, 6 8 and 12 hours after start of infusion
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: μg*h/mL
Arm/Group | Voriconazole IV
Number analyzed (Participants) | 25
μg*h/mL
  Day 1 | 21.18 (6.80)
  Day 7 (up to Day 20) | 36.21 (9.20)

12. Secondary Outcome: Cmax,ss of N-oxide Voriconazole Metabolite (UK-121, 265) Following IV Administration
Time Frame: as for outcome 11
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: μg/mL
Arm/Group | Voriconazole IV
Number analyzed (Participants) | 25
μg/mL
  Day 1 | 2.50 (0.84)
  Day 7 (up to Day 20) | 3.48 (0.73)

13. Secondary Outcome: Tmax of N-oxide Voriconazole Metabolite (UK-121, 265) Following IV Administration
Time Frame: as for outcome 11
Population: as for outcome 2
Measure: Median (Full Range); unit: μg*h/mL
Arm/Group | Voriconazole IV
Number analyzed (Participants) | 25
μg*h/mL
  Day 1 | 4.00 [1.97 to 8.03]
  Day 7 (up to Day 20) | 4.03 [0.00 to 12.10]

14. Secondary Outcome: AUC12,ss of N-oxide Voriconazole Metabolite (UK-121, 265) Following Oral Administration
Description: as for outcome 1
Time Frame: On Day 7 (up to Day 30) at predose, 1, 2, 4, 6, 8, and 12 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: μg*h/mL
Arm/Group | Voriconazole Oral
Number analyzed (Participants) | 19
μg*h/mL | 44.07 (13.86)

15. Secondary Outcome: Cmax,ss of N-oxide Voriconazole Metabolite (UK-121, 265) Following Oral Administration
Time Frame: Day 7 (up to Day 30) at predose, 1, 2, 4, 6, 8, and 12 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: μg/mL
Arm/Group | Voriconazole Oral
Number analyzed (Participants) | 19
μg/mL | 4.44 (1.43)

16. Secondary Outcome: Tmax of N-oxide Voriconazole Metabolite (UK-121, 265) Following Oral Administration
Time Frame: Day 7 (up to Day 30) at predose, 1, 2, 4, 6, 8, and 12 hours postdose
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Voriconazole Oral
Number analyzed (Participants) | 19
hours | 5.97 [1.00 to 8.10]

17. Other Pre Specified Outcome: Pharmacokinetic Parameters of Voriconazole in Adolescents Compared to Historical Adult Data - AUC12 IV Loading Dose.
Description: Data for this Outcome Measure are not reported here because the analysis population includes participants who were not enrolled in this study. ClinicalTrials.gov is designed for reporting results from only those participants who were enrolled in the study and described in the Participant Flow and Baseline Characteristics modules.
Time Frame: Day 1
Reporting Status: Not Posted
Measure: Geometric Mean (Full Range); unit: mcg*hr/mL

18. Other Pre Specified Outcome: Pharmacokinetic Parameters of Voriconazole in Adolescents Compared to Historical Adult Data - AUC12 IV Steady State
Description: as for outcome 17
Time Frame: Day 7 of IV dosing
Reporting Status: Not Posted
Measure: Geometric Mean (Full Range); unit: mcg*hr/mL

19. Other Pre Specified Outcome: Pharmacokinetic Parameters of Voriconazole in Adolescents Compared to Historical Adult Data - AUC12 Oral Dose All Subjects
Description: as for outcome 17
Time Frame: Day 7 Oral dosing
Reporting Status: Not Posted
Measure: Geometric Mean (Full Range); unit: mcg*hr/mL

20. Other Pre Specified Outcome: Pharmacokinetic Parameters of Voriconazole in Adolescents Compared to Historical Adult Data - AUC12 Oral 300mg
Description: as for outcome 17
Time Frame: Day 7 oral dosing
Reporting Status: Not Posted
Measure: Geometric Mean (Full Range); unit: mcg*hr/mL

21. Other Pre Specified Outcome: Pharmacokinetic Parameters of Voriconazole in Adolescents Compared to Historical Adult Data - Cmax IV Loading Dose
Description: as for outcome 17
Time Frame: Day 1
Reporting Status: Not Posted
Measure: Geometric Mean (Full Range); unit: mcg/mL

22. Other Pre Specified Outcome: Pharmacokinetic Parameters of Voriconazole in Adolescents Compared to Historical Adult Data - Cmax IV Steady State
Description: as for outcome 17
Time Frame: Day 7 of Intravenous dosing
Reporting Status: Not Posted
Measure: Geometric Mean (Full Range); unit: mcg/mL

23. Other Pre Specified Outcome: Pharmacokinetic Parameters of Voriconazole in Adolescents Compared to Historical Adult Data - Cmax Day 7 Oral All Participants
Description: as for outcome 17
Time Frame: Day 7 of oral dosing
Reporting Status: Not Posted
Measure: Geometric Mean (Full Range); unit: mcg/mL

24. Other Pre Specified Outcome: Pharmacokinetic Parameters of Voriconazole in Adolescents Compared to Historical Adult Data - Cmax 300 mg Oral Dose
Description: as for outcome 17
Time Frame: Day 7 of oral dosing
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Voriconazole IV | Voriconazole Oral
Serious Adverse Events (participants affected / at risk) | 4/26 | 4/22
Other Adverse Events (participants affected / at risk) | 26/26 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Voriconazole IV (N=26) | Voriconazole Oral (N=22)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Caecitis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Mucosal inflammation (General disorders) | 1 | 0
Acute graft versus host disease in intestine (Immune system disorders) | 0 | 1
Acute graft versus host disease in liver (Immune system disorders) | 0 | 1
Alpha haemolytic streptococcal infection (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Herpes simplex (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Capillary leak syndrome (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Voriconazole IV (N=26) | Voriconazole Oral (N=22)
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Coagulopathy (Blood and lymphatic system disorders) | 1 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 3 | 2
Pancytopenia (Blood and lymphatic system disorders) | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 3
Tachycardia (Cardiac disorders) | 1 | 0
Colour blindness (Congenital, familial and genetic disorders) | 0 | 1
Ear canal erythema (Ear and labyrinth disorders) | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 2
Conjunctival irritation (Eye disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 1 | 1
Conjunctivitis allergic (Eye disorders) | 1 | 1
Dry eye (Eye disorders) | 1 | 0
Hypermetropia (Eye disorders) | 0 | 1
Photophobia (Eye disorders) | 0 | 1
Strabismus (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 3
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2
Anorectal disorder (Gastrointestinal disorders) | 1 | 1
Ascites (Gastrointestinal disorders) | 1 | 2
Breath odour (Gastrointestinal disorders) | 1 | 1
Chapped lips (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 4
Diarrhoea (Gastrointestinal disorders) | 5 | 5
Dyspepsia (Gastrointestinal disorders) | 1 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 1
Faecal volume increased (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 1
Gingival bleeding (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 2 | 3
Haematochezia (Gastrointestinal disorders) | 2 | 3
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Lip dry (Gastrointestinal disorders) | 1 | 0
Lip haemorrhage (Gastrointestinal disorders) | 1 | 0
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 1 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 6 | 6
Oral pain (Gastrointestinal disorders) | 3 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Rectal fissure (Gastrointestinal disorders) | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 0
Toothache (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 5 | 5
Catheter related complication (General disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Chills (General disorders) | 1 | 2
Drug withdrawal syndrome (General disorders) | 0 | 1
Face oedema (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 2
Gait disturbance (General disorders) | 0 | 1
Generalised oedema (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 11 | 9
Oedema (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 4
Pain (General disorders) | 2 | 2
Pyrexia (General disorders) | 13 | 5
Suprapubic pain (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 1
Hepatomegaly (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 4 | 3
Jaundice (Hepatobiliary disorders) | 1 | 0
Acute graft versus host disease in intestine (Immune system disorders) | 0 | 1
Acute graft versus host disease in skin (Immune system disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Engraftment syndrome (Immune system disorders) | 3 | 1
Graft versus host disease (Immune system disorders) | 1 | 3
Hypogammaglobulinaemia (Immune system disorders) | 1 | 1
Adenovirus infection (Infections and infestations) | 1 | 0
BK virus infection (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 2 | 2
Bacterial infection (Infections and infestations) | 0 | 1
Catheter related infection (Infections and infestations) | 0 | 1
Cellulitis orbital (Infections and infestations) | 1 | 1
Central line infection (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 3
Cytomegalovirus viraemia (Infections and infestations) | 0 | 2
Escherichia bacteraemia (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 1 | 1
Human polyomavirus infection (Infections and infestations) | 1 | 1
Klebsiella bacteraemia (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 2
Oral herpes (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 0 | 1
Pneumonia fungal (Infections and infestations) | 0 | 2
Sinusitis (Infections and infestations) | 1 | 3
Staphylococcal bacteraemia (Infections and infestations) | 1 | 2
Staphylococcal infection (Infections and infestations) | 0 | 1
Streptococcal bacteraemia (Infections and infestations) | 3 | 1
Streptococcal sepsis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urethritis (Infections and infestations) | 0 | 1
Varicella (Infections and infestations) | 1 | 1
Ear abrasion (Injury, poisoning and procedural complications) | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 | 1
Refractoriness to platelet transfusion (Injury, poisoning and procedural complications) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Blood bilirubin increased (Investigations) | 2 | 2
Blood cortisol decreased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 2 | 2
Blood pressure systolic increased (Investigations) | 1 | 1
Blood triglycerides increased (Investigations) | 0 | 1
Blood urea increased (Investigations) | 2 | 1
Breath sounds abnormal (Investigations) | 0 | 1
CSF protein increased (Investigations) | 0 | 1
Cardiac function test abnormal (Investigations) | 1 | 1
Cytomegalovirus test positive (Investigations) | 1 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 1
Hepatic enzyme increased (Investigations) | 3 | 3
Immunosuppressant drug level increased (Investigations) | 1 | 1
Oxygen saturation decreased (Investigations) | 1 | 5
Transaminases increased (Investigations) | 1 | 2
Virus urine test positive (Investigations) | 0 | 2
Weight decreased (Investigations) | 1 | 1
White blood cell count increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 3
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 2
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 4 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 5
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 5
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Burning sensation (Nervous system disorders) | 0 | 2
Dizziness (Nervous system disorders) | 0 | 1
Drooling (Nervous system disorders) | 0 | 1
Dystonia (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 4 | 3
Mental impairment (Nervous system disorders) | 1 | 0
Myoclonus (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 1
Nystagmus (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 0
Sedation (Nervous system disorders) | 1 | 1
Tremor (Nervous system disorders) | 1 | 0
Agitation (Psychiatric disorders) | 0 | 2
Confusional state (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 1
Drug dependence (Psychiatric disorders) | 0 | 1
Flat affect (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 3
Mental status changes (Psychiatric disorders) | 0 | 1
Nightmare (Psychiatric disorders) | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 2
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 6
Glycosuria (Renal and urinary disorders) | 1 | 1
Haematuria (Renal and urinary disorders) | 3 | 5
Ketonuria (Renal and urinary disorders) | 2 | 1
Micturition disorder (Renal and urinary disorders) | 0 | 1
Oliguria (Renal and urinary disorders) | 2 | 1
Proteinuria (Renal and urinary disorders) | 2 | 2
Renal impairment (Renal and urinary disorders) | 2 | 2
Urinary retention (Renal and urinary disorders) | 0 | 1
Perineal pain (Reproductive system and breast disorders) | 0 | 1
Pruritus genital (Reproductive system and breast disorders) | 1 | 1
Scrotal pain (Reproductive system and breast disorders) | 1 | 1
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 2
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1
Purpura (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 4 | 5
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 3
Rash morbilliform (Skin and subcutaneous tissue disorders) | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Refusal of treatment by patient (Social circumstances) | 0 | 1
Oxygen supplementation (Surgical and medical procedures) | 0 | 1
Capillary leak syndrome (Vascular disorders) | 0 | 1
Flushing (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 4 | 6
Hypotension (Vascular disorders) | 2 | 5
Vena cava thrombosis (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.